CLINICAL TRIAL: NCT06264128
Title: The Effect on Subjective Comfort of a Device Providing Positive Airway Pressure (PAP) Drops During Inspiration (TPAP) Compared to Continuous Positive Airway Pressure (CPAP) in Obstructive Sleep Apnea Patients
Brief Title: TPAP for Comfort in OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SleepRes Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TheraPAP Comfort
Record Dates: First submitted 2024-02-02; First posted 2024-02-16 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: CPAP; comfort
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: All participants will undergo the same therapy combinations. CPAP (Continuous Positive Airway Pressure) and 2 level of TPAP (TheraPAP - novel CPAP approach pressure is reduced below therapy pressure from inspiration through mid exhalation specifically for comfort) will be assessed against each other in a round robin both backward and forward (6 total binary comparisons) for 2 levels of baseline pressure.
Masking Description: There is no specific intent to mask although participants will be naive to CPAP-type therapy, but they will be able to feel the difference.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- CPAP v TPAP (Experimental): Participants will compare CPAP to 2 different levels of TPAP, then will compare 2 levels of TPAP against each other by breathing on each pair of therapies for a minute or so, then deciding which is more comfortable or if they are equivalent.
  Interventions: Device: TPAP; Device: CPAP

INTERVENTIONS:
Device: TPAP — TPAP is a form of CPAP therapy where the therapy pressure is reduced from the beginning of inhalation through mid or later exhalation. The "CPAP" therapy pressure is only present at the end of the expiratory phase.
Device: CPAP — CPAP is a standard formal at home therapy for obstructive sleep apnea where a device attached via a facemask applies a constant pressure to a patient's lungs during sleep. It is the reference standard in this study.

SUMMARY:
TheraPAP is a prototype device (with full documented electrical and isolation safety) being developed by SleepRes for the treatment of obstructive sleep apnea (OSA) that can deliver either standard CPAP at a set pressure or what is called TPAP . TPAP is a pressure control algorithm that lowers the pressure from the set pressure at the beginning of inspiration and does not return the pressure to the full set level until about halfway through expiration. The present study, TheraPAP Comfort, aims at assessing whether TPAP improves patient comfort vs. CPAP during supine wakefulness.

DETAILED DESCRIPTION:
The TheraPAP Comfort Study is an in-office study to assess comfort of TPAP vs. CPAP in CPAP-naïve patients with OSA during supine wakefulness. Patients will be recruited after routine outpatient visits. They will be asked to breath normally for approximately 1 minute in supine wakefulness while being administered background CPAP (at 9 or 13 cmH2O) or TPAP at various pressure drops. TPAP drops will be administered in a paired comparison before or/and after each corresponding CPAP level, according to a randomized design. Eventually, 6 one-to-one comparisons (TPAP vs. corresponding background CPAP or TPAP vs. TPAP) will be made, 3 per each randomized order. As an example, CPAP 9 will be compared to TPAP 1/1 cmH2O drops; CPAP 9 will be compared to TPAP 2/2 cmH2O drops; and TPAP 1/1 cmH2O drops will be compared to TPAP 2/2 cmH2O drops in a random sequence.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 70 age range
* AHI (apnea/hypopnea index) > 10 on a previous HST (Home Sleep Test)
* CPAP-naive participants
* BMI (Body Mass Index) >= 18 kg/m^2

Exclusion Criteria:

1. Current clinically significant sleep disorder other than OSA (Obstructive Sleep Apnea) of a severity that would interfere with study participation or interpretability of data (including central sleep apnea, per central AHI > 5 events/h).
2. Any chronic lung diseases.
3. Chronic oxygen therapy.
4. A serious illness or infection in the past 30 days as determined by investigator.
5. Patients with hypoglossal nerve stimulation implant.
6. Any non-previously mentioned vulnerable population.
7. Any condition that in the investigator's opinion would present an unreasonable risk to the participant, or which would interfere with their participation in the study or confound study interpretation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abinash Joshi, MD, Principal Investigator — University of Louisville
Locations (1):
- SleepCenters of Middle Tennessee, Murfreesboro, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
We only plan to share the results after we publish them.

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Period 1: CPAP Period 2: TPAP
  This was a trial in which the same participant underwent multiple testing in sequence and on the same session after being randomized only once (to CPAP or TPAP first). As such, only two sequences are present.
  CPAP was initially administered at 9 cmH2O TPAP was initially reduced by 2+2 cmH2O
  If the participant chose TPAP, the test was repeated as follows (see also below):
  CPAP was administered at 13 cmH2O TPAP was reduced by 2+3 cmH2O
  If the participant chose TPAP, testing ended.
  If the participant, instead, had chosen CPAP at 9 cmH2O, the test was repeated as follows:
  CPAP was administered at 9 cmH2O TPAP was reduced by 1+2 cmH2O
  If the participant chose TPAP, testing ended.
  If the participant chose CPAP at 9 cmH2O, the test was repeated as follows:
  CPAP was administered at 9 cmH2O TPAP was reduced by 1+1 cmH2O
  Regardless, of the choice, the testing was repeated as follows:
  CPAP was administered at 13 cmH2O TPAP was reduced by 2+3 cmH2O
  If the participant chose TPAP, testing ended.
  If the participant chose CPAP at 13 cmH2O, testing was repeated as follows:
  CPAP was administered at 13 cmH2O TPAP was reduced by 2+2 cmH2O
  If the participant chose TPAP, testing ended.
  If the participant chose CPAP at 13 cmH2O, testing was repeated as follows:
  CPAP was administered at 13 cmH2O TPAP was reduced by 1+2 cmH2O
  Regardless of choices, testing ended after this.
- Sequence 2: Period 1: TPAP Period 2: CPAP
  This was a trial in which the same participant underwent multiple testing in sequence and on the same session after being randomized only once (to CPAP or TPAP first). As such, only two sequences are present.
  TPAP was initially reduced by 2+2 cmH2O CPAP was initially administered at 9 cmH2O
  If the participant chose TPAP, the test was repeated as follows (see also below):
  TPAP was reduced by 2+3 cmH2O CPAP was administered at 13 cmH2O
  If the participant chose TPAP, testing ended.
  If the participant, instead, had chosen CPAP at 9 cmH2O, the test was repeated as follows:
  TPAP was reduced by 1+2 cmH2O CPAP was administered at 9 cmH2O
  If the participant chose TPAP, testing ended.
  If the participant chose CPAP at 9 cmH2O, the test was repeated as follows:
  TPAP was reduced by 1+1 cmH2O CPAP was administered at 9 cmH2O
  Regardless, of the choice, the testing was repeated as follows:
  TPAP was reduced by 2+3 cmH2O CPAP was administered at 13 cmH2O
  If the participant chose TPAP, testing ended.
  If the participant chose CPAP at 13 cmH2O, testing was repeated as follows:
  TPAP was reduced by 2+2 cmH2O CPAP was administered at 13 cmH2O
  If the participant chose TPAP, testing ended.
  If the participant chose CPAP at 13 cmH2O, testing was repeated as follows:
  TPAP was reduced by 1+2 cmH2O CPAP was administered at 13 cmH2O
  Regardless of choices, testing ended after this.
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2
Started | 74 | 76
Completed | 74 | 76
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Group: All participants in the study (who crossovered from one treatment arm to the other)
Arm/Group | Overall Group
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 123
  More than one race | 0
  Unknown or Not Reported | 7

OUTCOME MEASURES:

1. Primary Outcome: CPAP v TPAP Patient Preference at 9 cmH2O Baseline Pressure, TPAP Drop 2+2 cmH2O
Description: Compare the comfort level of CPAP at 9 cmH2O against TPAP dropped by 2+2 cmH2O
Time Frame: All tests conducted in a 20 minute time frame on awake supine patients.
Population: The outcome refers to % of participants who preferred TPAP over CPAP
Measure: Number (95% Confidence Interval); unit: percentage of total participants
Groups:
- CPAP vs. TPAP (Baseline Pressure: 9 cmH2O ): CPAP at 9 cmH2O TPAP at 9 cmH2O with sequential comfort drops of 2+2 cmH2O
Arm/Group | CPAP vs. TPAP (Baseline Pressure: 9 cmH2O )
Number analyzed (Participants) | 150
percentage of total participants | 69.3 [61 to 77]

2. Primary Outcome: CPAP v TPAP Patient Preference at 13 cmH2O Baseline Pressure, TPAP Drop 2+3 cmH2O
Description: Compare the comfort level of CPAP at 13 cmH2O against TPAP dropped by 2+3 cmH2O
Time Frame: All tests conducted in a 20 minute time frame on awake supine patients.
Population: The outcome refers to % of participants who preferred TPAP over CPAP
Measure: Number (95% Confidence Interval); unit: percentage of total participants
Groups:
- CPAP vs. TPAP (Baseline Pressure: 13 cmH2O ): CPAP at 13 cmH2O TPAP at 13 cmH2O with sequential comfort drops of 2+3 cmH2O
Arm/Group | CPAP vs. TPAP (Baseline Pressure: 13 cmH2O )
Number analyzed (Participants) | 150
percentage of total participants | 84 [77 to 89]

3. Secondary Outcome: CPAP v TPAP Patient Preference at 9 cmH2O Baseline Pressure, TPAP Drop 1+2 cmH2O
Time Frame: All tests conducted in a 20 minute time frame on awake supine patients.
Population: The outcome data refers to participants (N=21) who preferred TPAP (with a 1+2 cmH2O drop) over CPAP at 9 cmH2O. Notably, this was a repeated test among participants who initially did not prefer TPAP in the comparison between CPAP at 9 cmH2O and TPAP with a 2+2 cmH2O, independent of sequence. I.e., 46 participants found CPAP more comfortable than TPAP with 2+2 cmH2O drop, so testing continued with those individuals, of whom, eventually, 21 chose TPAP with 1+2 cmH2O drop.
Measure: Number; unit: percentage of total participants
Groups:
- CPAP vs. TPAP (Baseline Pressure: 9 cmH2O ): CPAP at 9 cmH2O TPAP at 9 cmH2O with sequential comfort drops of 1+2 cmH2O
Arm/Group | CPAP vs. TPAP (Baseline Pressure: 9 cmH2O )
Number analyzed (Participants) | 46
percentage of total participants | 45.6

4. Secondary Outcome: CPAP v TPAP Patient Preference at 9 cmH2O Baseline Pressure, TPAP Drop 1+1 cmH2O
Time Frame: All tests conducted in a 20 minute time frame on awake supine patients.
Population: The outcome data refers to participants (N=14) who preferred TPAP (with a 1+1 cmH2O drop) over CPAP at 9 cmH2O. Notably, this was a repeated test among participants who initially did not prefer TPAP in the comparison between CPAP at 9 cmH2O and TPAP with a 2+2 cmH2O or with at 1+2 cmH2O drop, independent of sequence. I.e., only 25 participants found CPAP more comfortable than TPAP at any drop, so testing continued with those individuals, of whom, eventually, 14 chose TPAP with 1+1 cmH2O drop.
Measure: Number; unit: percentage of total participants
Groups:
- CPAP vs. TPAP (Baseline Pressure: 9 cmH2O ): CPAP at 9 cmH2O TPAP at 9 cmH2O with sequential comfort drops of 1+1 cmH2O
Arm/Group | CPAP vs. TPAP (Baseline Pressure: 9 cmH2O )
Number analyzed (Participants) | 25
percentage of total participants | 56

5. Secondary Outcome: CPAP v TPAP Patient Preference at 13 cmH2O Baseline Pressure, TPAP Drop 2+2 cmH2O
Time Frame: All tests conducted in a 20 minute time frame on awake supine patients.
Population: The outcome data refers to participants (N=11) who preferred TPAP (with a 2+2 cmH2O drop) over CPAP at 13 cmH2O. Notably, this was a repeated test among participants who initially did not prefer TPAP in the comparison between CPAP at 13 cmH2O and TPAP with a 2+3 cmH2O, independent of sequence. I.e., only 24 participants found CPAP more comfortable than TPAP with 2+3 cmH2O drop, so testing continued with those individuals, of whom, eventually, 11 chose TPAP with 2+2 cmH2O drop.
Measure: Number; unit: percentage of total participants
Groups:
- CPAP vs. TPAP (Baseline Pressure: 13 cmH2O ): CPAP at 13 cmH2O TPAP at 13 cmH2O with sequential comfort drops of 2+2 cmH2O
Arm/Group | CPAP vs. TPAP (Baseline Pressure: 13 cmH2O )
Number analyzed (Participants) | 24
percentage of total participants | 45.8

6. Secondary Outcome: CPAP v TPAP Patient Preference at 13 cmH2O Baseline Pressure, TPAP Drop 1+2 cmH2O
Time Frame: All tests conducted in a 20 minute time frame on awake supine patients.
Population: The outcome data refers to participants (N=5) who preferred TPAP (with a 1+2 cmH2O drop) over CPAP at 13 cmH2O.Notably, this was a repeated test among participants who initially did not prefer TPAP in the comparison between CPAP at 13 cmH2O and TPAP with a 2+3 cmH2O or with at 2+2 cmH2O drop, independent of sequence. I.e., only 13 participants found CPAP more comfortable than TPAP at any drop, so testing continued with those individuals, of whom, eventually, 5 chose TPAP with 1+2 cmH2O drop
Measure: Number; unit: percentage of total participants
Groups:
- CPAP vs. TPAP (Baseline Pressure: 13 cmH2O ): CPAP at 13 cmH2O TPAP at 13 cmH2O with sequential comfort drops of 1+2 cmH2O
Arm/Group | CPAP vs. TPAP (Baseline Pressure: 13 cmH2O )
Number analyzed (Participants) | 13
percentage of total participants | 38.5

ADVERSE EVENTS:
Time Frame: 20 minute office visit
Groups:
- TPAP: TPAP group at baseline pressure of 9 or 13 cmH2O. Testing was done in series within the same sequence
- CPAP: CPAP group at baseline pressure of 9 or 13 cmH2O. Testing was done in series within the same sequence
Arm/Group | TPAP | CPAP
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/150
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/150
Other Adverse Events (participants affected / at risk) | 0/150 | 0/150

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT06264128/Prot_SAP_001.pdf